CLINICAL TRIAL: NCT05369208
Title: An Open-label Study to Evaluate the Efficacy and Safety of Avatrombopag for the Treatment of Thrombocytopenia in Japanese Adults With Chronic Immune Thrombocytopenia
Brief Title: Evaluation of Avatrombopag for the Treatment of Thrombocytopenia in Japanese Adults With Chronic ITP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA-ITP-307
Record Dates: First submitted 2022-04-21; First posted 2022-05-11 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Avatrombopag (Other): Avatrombopag 20 mg oral tablet
  Interventions: Drug: Avatrombopag Oral Tablet

INTERVENTIONS:
Drug: Avatrombopag Oral Tablet — Avatrombopag 20 mg given once daily (initial dose). Dosage adjustments were determined by the physician to maintain a platelet count between 50 x 10^9 to 200 x 10^9 as defined in the protocol and in accordance with overseas labeling.
  Other Names: Doptelet

SUMMARY:
Evaluate the efficacy, safety, and PK of avatrombopag given for 26 weeks in Japanese adults with chronic immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
This Phase 3, multicenter, open label study will evaluate the efficacy, safety, and population pharmacokinetics (PK) of avatrombopag in Japanese adults with chronic ITP. At least 19 subjects will be enrolled. The study will consist of 3 phases: Pre-enrollment, Primary Investigation, and Extension Phase until market authorization in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of chronic immune thrombocytopenia (ITP) (≥12 months duration) and has had an insufficient response to a previous ITP treatment, in the opinion of the Investigator.
* Subject has an average of 2 platelet counts <30×10^9/L (no single count can be >35×10^9/L). The 2 samples must be obtained ≥48 hours and ≤2 weeks apart.

Exclusion Criteria:

* Subjects with known secondary immune thrombocytopenia (e.g., with known Helicobacter pylori-induced ITP, subjects infected with known human immunodeficiency virus (HIV) or hepatitis C virus (HCV) or subjects with known systemic lupus erythematosus).
* Subjects with known inherited thrombocytopenia (e.g., Myosin Heavy Chain 9 (MYH-9) disorders) or hereditary thrombophilic disorders (e.g., Factor V Leiden, antithrombin III deficiency).
* History of myelodysplastic syndrome (MDS).
* History of arterial or venous thrombosis.
* Subjects with a history of significant cardiovascular disease (e.g., congestive heart failure (CHF) New York Heart Association Grade III/IV, arrhythmia known to increase the risk of thromboembolic events [e.g., atrial fibrillation], angina, coronary artery stent placement, angioplasty, coronary artery bypass grafting).
* Subjects with a history of cirrhosis, portal hypertension, or chronic active hepatitis.
* Subjects with concurrent malignant disease or receiving cytotoxic chemotherapy for a reason other than ITP treatment.
* Use of immunoglobulins (IVIg and anti-D) or corticosteroid rescue therapy within 1 week of Day 1/Baseline.
* Splenectomy or use of rituximab within 12 weeks of Day 1/Baseline.
* Use of romiplostim or eltrombopag within 1 week of Day 1/Baseline.
* Use of chronic corticosteroid treatment or azathioprine within 4 weeks of Day 1/Baseline, unless receiving a stable dose for at least 4 weeks.
* Use of mycophenolate mofetil, cyclosporin A, or danazol within 4 weeks of Day 1/Baseline, unless receiving a stable dose for at least 12 weeks.
* Use of cyclophosphamide or vinca alkaloid regimens within 4 weeks of Baseline Visit.
* Currently receiving moderate or strong dual inhibitors/inducers of CYP2C9 and CYP3A4.
* Serum creatinine ≥1.5× the upper limit of normal (ULN).
* Serum bilirubin ≥2×ULN.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3×ULN.
* Females who are pregnant (positive beta-human chorionic gonadotropin (β-hCG) test) or breastfeeding.
* Received treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) before Day 1/Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2025-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Japan (19):
  - Sobi Site 105, Toyohashi, Aichi-ken
  - Sobi Site 110, Tōon, Ehime
  - Sobi Site 118, Iizuka-shi, Fukuoka
  - Sobi Site 116, Kitakyushu, Fukuoka
  - Sobi Site 117, Kurume, Fukuoka
  - Sobi Site 114, Gifu, Gifu
  - Sobi Site 115, Fukuyama-shi, Hiroshima
  - Sobi Site 109, Hiroshima, Hiroshima
  - Sobi Site 108, Kobe, Hyōgo
  - Sobi Site 113, Kanazawa, Ishikawa-ken
  - Sobi Site 101, Shiwa-gun, Iwata
  - Sobi Site 111, Fujisawa, Kanagawa
  - Sobi Site 119, Kumamoto, Kumamoto
  - Sobi Site 107, Hirakata, Osaka
  - Sobi Site 106, Suita, Osaka
  - Sobi Site 104, Hachiōji-shi, Tokyo
  - Sobi Site 103, Bunkyō City, Toyko
  - Sobi Site 102, Chuo-shi, Yamanashi
  - Sobi Site 112, Kofu, Yamanashi

RESULTS

PARTICIPANT FLOW:
Groups:
- Avatrombopag: Avatrombopag 20 mg oral tablet
  Avatrombopag 20 mg given once daily (initial dose). Dosage adjustments were determined by the physician to maintain a platelet count between 50 x 10^9 to 200 x 10^9 as defined in the protocol and in accordance with overseas labeling.
Period: Core Phase
Arm/Group | Avatrombopag
Started | 19
Completed | 15
Not Completed | 4
Not completed — Prohibited Medication Required | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Period: Extension Phase
Arm/Group | Avatrombopag
Started | 15
Completed | 0
Not Completed | 15

BASELINE CHARACTERISTICS:
Groups:
- Avatrombopag: Avatrombopag 20 mg oral tablet
  Avatrombopag 20 mg given once daily (initial dose). Dose adjustments were determined by the physician to maintain a platelet count between 50 x 10^9 to 200 x 10^9 as defined in the protocol and in accordance with the overseas labeling.
Arm/Group | Avatrombopag
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (16.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 19

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Number of Weeks of Platelet Response
Description: Cumulative number of weeks in which the platelet count is ≥50×10^9/L during 26 weeks of treatment in the absence of rescue therapy.
Time Frame: 26 weeks of active treatment
Population: Full analysis set of core phase
Measure: Mean (Standard Deviation); unit: cumulative number of weeks
Arm/Group | Avatrombopag
Number analyzed (Participants) | 19
cumulative number of weeks | 13.47 (9.002)

2. Secondary Outcome: Response Rate at Day 8
Description: Proportion of subjects with a platelet response ≥50×10^9/L at Day 8 in the absence of rescue therapy
Time Frame: Day 8
Population: Full analysis set of core phase
Measure: Count of Participants; unit: Participants
Arm/Group | Avatrombopag
Number analyzed (Participants) | 19
Participants | 12

ADVERSE EVENTS:
Time Frame: Up to 26 weeks of treatment and a 4 week follow up period (Core Phase)
Description: Avatrombopag reported as a single group. Adverse events were not grouped by dose since the dosage regimen could be adjusted frequently throughout the study.
Arm/Group | Avatrombopag
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 3/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avatrombopag (N=19)
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 (1)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avatrombopag (N=19)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Scleral Haemorrhage (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Tooth Fracture (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bacterial Infection (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
Chronic Sinusitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1)
Blood Pressure Decreased (Investigations) | 1 (1)
Blood Pressure Increased (Investigations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3)
Hypotension (Vascular disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are not allowed to publish clinical trial data on their own after trial completion.

DOCUMENTS (2):
  • Study Protocol (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT05369208/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT05369208/SAP_001.pdf